CLINICAL TRIAL: NCT02326441
Title: A Phase 1 Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetics of KX2-361 in Subjects With Advanced Malignancies That Are Refractory to Conventional Therapies
Brief Title: Safety, Tolerability & PK of KX2-361 in Subjects w Adv. Malignancies Refractory to Conventional Therapies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Athenex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KX02-01-13
Record Dates: First submitted 2014-12-10; First posted 2014-12-29 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Advance Malignancies
Keywords: advanced malignancies; refractory therapies; phase 1
MeSH Terms: interventions — KX2-361

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- KX2-361 (Experimental)
  Interventions: Drug: KX2-361

INTERVENTIONS:
Drug: KX2-361

SUMMARY:
The purpose of this study is to determine the safety and tolerability of the study drug KX2-361 and to determine how much of the study drug enters the bloodstream, in patients with advanced malignancies that have not responded to conventional therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. Adults ≥ 18 years of age.
3. Dose Escalation Cohort only:

   Confirmed advanced solid tumor or lymphoma for which standard curative or palliative measures do not exist or are no longer effective; subjects with progressive brain metastases are also eligible.

   OR Confirmed Histological/cytological hematological malignancy that is refractory to/relapsed after and/or intolerant of standard therapies or for which no standard therapy exists.

   OR Confirmed high grade glioma (grade 3and4) that is relapsed/refractory to standard therapies and who have progressive disease following radiation therapy. Patients with any number of prior treatments are allowed.
   * Expansion Cohort only:

   Patients with high grade glioma (grade 3 and 4) that are refractory to standard therapies, and who have progressive disease following radiation therapy. Patients with any number of prior treatments are allowed.
4. ECOG performance status of 0-2, Karnofsky Performance Status ≥60 (for glioma subjects).
5. Life expectancy of at least 12 weeks.
6. The following laboratory values:

   * ANC ≥ 1.5 x 10⁹/L
   * Platelets ≥ 100 x 10⁹/L
   * Hemoglobin (Hgb) > 10 g/dL
   * Serum total bilirubin ≤ 1.5 x ULN
   * ALT and AST ≤ 3.0 x ULN (subjects with known liver metastases may have AST and ALT ≤ 5.0 x ULN)
   * Serum creatinine ≤ 1.5 x ULN or calculated creatinine clearance (using Cockcroft and Gault method) > 60 mL/min)
7. Willingness to use acceptable birth control. Subjects with the potential for pregnancy or impregnating their partner must agree to follow acceptable birth control methods to avoid conception. Female subjects of child-bearing potential must have a negative pregnancy test.

Exclusion Criteria:

1. Subjects who have not recovered to Grade 0 or 1 toxicity from previous anti-cancer treatments or previous investigational agents.
2. Subjects who have received investigational agents within 28 days of the first day of study drug.
3. Subjects with primary CNS malignancy other than high grade glioma (Grade 3 or 4)
4. Subjects who have received extensive radiation therapy, including sternum, pelvis, scapulae, vertebrae or skull, within 4 weeks of the first day of study drug or received palliative low dose radiation therapy limited to limbs within 1 week of the first day of study drug, or subjects who have not recovered from side effects of such therapy.
5. Subjects who are currently taking or have received hormones (eg, estrogen or progesterone) within 7 days the first dose of study drug. Note: Luteinizing hormone-releasing hormone (LHRH) analogs are permissible.
6. Subjects who are using moderate or strong CYP450 3A4 modulators (with the exception of antifungal agents listed in Appendix 2) within 5 half-lives before the first dose of study drug.
7. Subjects who are using prescription or OTC medications (including, for example, proton pump inhibitors, H2 antagonists or calcium carbonate) that reduce or neutralize gastric acidity within 5 half lives before the first dose of study drug. Use of these medications for supportive care after cycle 1 is permitted.
8. Subjects who had major surgery within 4 weeks of the first day of study drug.
9. Subjects who had major surgery to the upper gastrointestinal tract, or who have a history of inflammatory bowel disease, malabsorption syndrome, or other medical condition that may interfere with oral drug absorption.
10. Subjects with a history of intestinal perforation, colitis, clinically significant gastrointestinal bleeding or intestinal obstruction within one year prior to enrollment.
11. Subjects with signs or symptoms of other major diseases including, but not limited to: end organ failure, major chronic illnesses other than cancer, coagulation disorders, hemolytic conditions (eg, sickle cell disease ) or active infections that, in the opinion of the investigator, make it undesirable for the subject to participate in the study.
12. Subjects who have a history of major cardiac or neurologic disease including, but not limited to, angina pectoris, symptomatic coronary artery disease, uncontrolled hypertension (at time of study entry), New York Heart Association (NYHA) Class III or IV congestive heart failure, confirmed significant cardiac conduction abnormalities (including QTc > 0.45 sec) or arrhythmias, myocardial infarction within 12 months, cerebrovascular accidents, or transient ischemic attacks.
13. Other conditions which could jeopardize the subject's ability to comply with the protocol including but not limited to dementia, psychosis, or other major psychiatric disorder.
14. Subjects with a known history of hepatitis B or C or human immunodeficiency (HIV) infection.
15. Subjects who require therapeutic doses of anticoagulants.
16. Subjects who require the use of granulocyte colony stimulating factors (GCSF) for prophylaxis of neutropenia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-12; Primary Completion 2017-07 (Actual); Study Completion 2018-05-23 (Actual)

PRIMARY OUTCOMES:
Define MTD | 12 months
  The Maximum Tolerated Dose is defined as one dose level below where two or more subjects experienced a dose limiting toxicity (DLT).

SECONDARY OUTCOMES:
Safety and Tolerability assessed by adverse events and changes in laboratory parameters | 24 months
  Patient incidence of adverse events will be displayed by dose group and by system organ class. Adverse events will also be summarized by severity and relationship to the study drug. Laboratory parameters assessed will include vital signs, history and PE, assessment of toxicity, complete blood count w differentials and reticulocytes, serum chemistry (incl. RDB, LFT serum amylase and serum lipase), PT (or INR/PTT), urinalysis, and ECG assessment.
Pharmacokinetics (rofile pharmacokinetic outcome measures, e.g. Cmax, Tmax, AUCt, AUC0-inf, t½, CL, and Css) | 24 months
  Plasma concentrations of KX2-361 will be analyzed to determine profile pharmacokinetic outcome measures, e.g. Cmax, Tmax, AUCt, AUC0-inf, t½, CL, and Css etc.
Activity in escalation and expansion cohorts (according to the RECIST criteria, CHESON criteria, or the Modified RANO) | 24 months
  Activity response for the Dose Escalation Cohort portion of the study will be assessed by the investigator according to the RECIST criteria, CHESON criteria, or the Modified RANO criteria. The Expansion Cohort will utilize the Modified RANO criteria only for response measurements.

CONTACTS AND LOCATIONS:
Overall Officials: David Cutler, MD, Study Director — Kinex Pharmaceutical
Locations (3):
- United States (3):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Cleveland Clinic, Taussig Cancer Institute, Cleveland, Ohio
  - UTHSCSA Cancer Therapy and Research Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided